CLINICAL TRIAL: NCT04816149
Title: Development of a Novel Couples-Based Suicide Intervention: Treatment for Relationships and Safety Together (TR&ST)
Brief Title: Treatment for Relationships and Safety Together
Acronym: TR&ST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3490-W; RX003490 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2021-03-17; First posted 2021-03-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Suicide; Interpersonal Relations
Keywords: Suicide; Interpersonal Relations
MeSH Terms: conditions — Suicide | interventions — Therapeutics; Association

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VA Standard Suicide Intervention (Active Comparator): Our active control condition is standardized and contains the elements of standard practice suicide-specific intervention delivered at the VA, which include: 1) suicide risk assessment using the CSSR-S, 2) VA Safety Planning Intervention, 3) timely referral to VA mental health outpatient care, including couples intervention (engagement will be tracked), and 4) Suicide Prevention Coordinator (SPC) follow-up contacts (which have been found to significantly reduce suicidal behavior).
  Interventions: Behavioral: VA Standard Suicide Intervention
- Treatment for Relationships and Safety Together (TR&ST) (Experimental): TR&ST consists of eleven 90-minute sessions delivered in three phases. During phase one, couples receive a tailored cognitive-behavioral conceptualization of suicide and relationship distress based on clinical interview, as well as psychoeducation about their bidirectional influences. They also engage in behavioral activation focused on positive couple activities, emotion regulation, distress tolerance, and conflict management strategies. In phase two, couples learn communication skills and discuss suicidal thoughts and behaviors, as well as their relationship challenges that interact with suicidal thoughts and behavior. Phase three is focused on conjoint thought challenging to shift dysfunctional cognitions related to suicide and relationship problems.
  Interventions: Behavioral: Treatment for Relationships and Safety Together (TR&ST)

INTERVENTIONS:
Behavioral: VA Standard Suicide Intervention — Our active control condition is standardized and contains the elements of standard practice suicide-specific intervention delivered at the VA, which include: 1) suicide risk assessment using the CSSR-S, 2) VA Safety Planning Intervention, 3) timely referral to VA mental health outpatient care, including couples intervention (engagement will be tracked), and 4) Suicide Prevention Coordinator (SPC) follow-up contacts (which have been found to significantly reduce suicidal behavior).
  Arms: VA Standard Suicide Intervention
Behavioral: Treatment for Relationships and Safety Together (TR&ST) — TR&ST consists of eleven 90-minute sessions delivered in three phases. During phase one, couples receive a tailored cognitive-behavioral conceptualization of suicide and relationship distress based on clinical interview, as well as psychoeducation about their bidirectional influences. They also engage in behavioral activation focused on positive couple activities, emotion regulation, distress tolerance, and conflict management strategies. In phase two, couples learn communication skills and discuss suicidal thoughts and behaviors, as well as their relationship challenges that interact with suicidal thoughts and behavior. Phase three is focused on conjoint thought challenging to shift dysfunctional cognitions related to suicide and relationship problems.
  Arms: Treatment for Relationships and Safety Together (TR&ST)

SUMMARY:
Suicide prevention is the top clinical priority for VA/DoD. Suicide is one of the leading causes of death in the United States and worldwide with suicide rates among U.S. military Veterans doubling (27.7 per 100,000) the rate of civilian levels. Despite a rise in prevention efforts, rates have continued to increase. Theories of suicide and rehabilitation psychology stress the importance of the person-environment interaction in contributing to one's disability experience. Several studies have found that the most frequent situation precipitating suicide was a problem with a romantic partner. In contrast, people with higher relationship satisfaction are less likely to have suicidal thoughts. Prevention of suicide in high risk Veterans is of vital importance and the quality of one's intimate relationship is an understudied intervention target for suicide prevention. Despite the fact that VA/DoD recommend and Veterans desire treatments that involve family members, currently no couple-based suicide-specific interventions exist. The goals of this CDA-II proposal are to refine and pilot a novel suicide-specific couple-based intervention: Treatment for Relationships and Safety Together (TR&ST). TR&ST adapts an evidence-based intervention for suicide, Brief Cognitive Behavioral Therapy (BCBT) for Suicide, to be dyadically focused and integrates Cognitive Behavioral Couple Therapy (CBCT) skills. The proposed 5-year study consists of two phases. Phase 1: treatment refinement with 12 couples (N=24) and Phase 2: pilot Randomized Controlled Trial (RCT) of TR&ST compared to VA Standard Suicide Intervention, which will involve suicide risk assessment, VA safety planning, Suicide Prevention Coordinator (SPC) follow-up, and referral to outpatient mental health with 60 couples (N=120). The intervention period is 11-weeks and the entire study period is approximately 7 months. Couples in both phases will be quantitatively assessed at baseline, mid-treatment, post-treatment, and 3-months post-treatment. The primary outcome to be evaluated is change in severity of suicidal thoughts. Secondary outcomes concern changes in interpersonal functioning theorized to influence suicidal thoughts and behavior.

DETAILED DESCRIPTION:
Suicide prevention is the top clinical priority for VA/DoD. Suicide is one of the leading causes of death in the United States and worldwide with suicide rates among U.S. military Veterans doubling (27.7 per 100,000) the rate of civilian levels. Despite a rise in prevention efforts, rates have continued to increase. Theories of suicide and rehabilitation psychology stress the importance of the person-environment interaction in contributing to one's disability experience. Several studies have found that the most frequent situation precipitating suicide was a problem with a romantic partner. In contrast, people with higher relationship satisfaction are less likely to have suicidal thoughts. The International Classification of Functioning, Disability and Health (ICF) identifies social engagement and communication as important components of functioning. Prevention of suicide in at-risk Veterans is of vital importance and the quality of one's intimate relationship is an understudied intervention target for suicide prevention. The importance of including family members in Veterans' suicide related care is a critical component of the National Strategy for Preventing Veteran Suicides 2018-2028, the National Action Alliance on Suicide Prevention, and a key finding from VA/DoD patient focus groups conducted for the 2019 VA/DoD Clinical Practice Guidelines for the Assessment and Management of Patients at Risk for Suicide. Despite the fact that VA/DoD recommend and Veterans desire treatments that involve family members, currently no couple-based suicide-specific interventions exist. The goals of this CDA-II are to refine and pilot a novel suicide-specific couple-based intervention-Treatment for Relationships and Safety Together (TR&ST). TR&ST adapts an evidence-based intervention for suicide, Brief Cognitive Behavioral Therapy (BCBT) for Suicide, to be dyadically focused and integrates Cognitive Behavioral Couple Therapy (CBCT) skills.

The proposed 5-year study consists of two phases. Phase 1: treatment refinement with 12 couples (N=24) and Phase 2: pilot Randomized Controlled Trial (RCT) of TR&ST compared to VA Standard Suicide Intervention, which will involve suicide risk assessment, VA safety planning, Suicide Prevention Coordinator (SPC) follow-up, and referral to outpatient mental health with 60 couples (N=120). The intervention period is 11-weeks and the entire study period is approximately 7 months. Couples in both phases will be quantitatively assessed at baseline, mid-treatment, post-treatment, and 3-months post-treatment. The primary outcome to be evaluated is change in severity of suicidal ideation. Secondary outcomes concern changes in interpersonal functioning theorized to influence suicidal ideation and behavior.

The Specific Aims of the study are:

Aim 1 (Phase 1): refine TR&ST in a population of Veterans with active suicidal ideation Aim 2 (Phase 2): evaluate feasibility and acceptability of TR&ST Hypothesis 1 is that TR&ST will be feasible to deliver, as evidenced by attainment of recruitment goals, retention rates 70%, and high credibility and expectancy ratings and satisfaction.

Aim 3 (Phase 2): estimate the preliminary impact of TR&ST vs. VA Standard Suicide Intervention on suicidal ideation severity and proximal targets of interpersonal functioning over 7 months to determine if a future efficacy trial is warranted.

Hypothesis 2a is that Veterans engaged in TR&ST (vs. VA Standard Suicide Intervention) will have greater reduction in suicidal ideation severity (primary outcome) Hypothesis 2b is that Veterans and partners engaged in TR&ST (vs. VA Standard Suicide Intervention) will have improved interpersonal functioning (i.e., communication, bonding, relationship satisfaction) Hypothesis 2c is that the effect of TR&ST on Veteran's reduced suicidal ideation will be mediated by improvements in Veteran and partner interpersonal functioning Exploratory Aim 1: examine rates of suicide related behavior for Veterans in TR&ST (vs. VA Standard Suicide Intervention) Exploratory Aim 2: examine links between weekly changes in suicidal ideation and relationship quality Exploratory Aim 3: examine the impact of TR&ST on depression, PTSD, and relationship conflict

ELIGIBILITY:
Inclusion Criteria:

* Veterans who report present suicidal ideation CSSR-S > 2 ("Active thoughts of killing oneself") in past 1 month at phone screen and/or a suicide attempt in the prior 3 months, and
* an intimate partner who is willing to participate.
* Additional inclusion criteria for both Veterans and Partners include:

  * in the committed relationship for at least 6 months
  * plans to remain in the San Diego region for 7 months
  * capable of informed consent
  * agree to have assessment and treatment sessions audio recorded.

Exclusion Criteria:

The following are our Exclusion Criteria for both Veterans and Partners:

* not English speaking
* cannot complete the assessment battery
* current substance use requiring immediate detoxification or outpatient plan directed specifically to residential substance use disorder (not mental health) services
* has or meets criteria for a current diagnosis of psychosis and/or mania in either member of the couple
* under conservatorship requiring proxy consent
* any perpetration of severe physical or sexual relationship aggression in the past year (as assessed by the CTS-2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in severity of suicidal ideation from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Beck Scale for Suicidal Ideation has a minimum possible score of 0, and maximum possible score of 38, wherein higher scores reflect more severe suicidal ideation.

SECONDARY OUTCOMES:
Change in positive communication from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Communication Skills Test has a minimum possible score of 10, and maximum possible score of 70, wherein higher scores reflect more positive communication.
Change in negative communication from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Communication Danger Signs Scale has a minimum possible score of 5, and maximum possible score of 15, wherein higher scores reflect more negative communication.
Change in positive bonding from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Positive Bonding Scale has a minimum possible score of 9, and maximum possible score of 63, wherein higher scores reflect more positive bonding.
Change in perceived burdensomeness and thwarted belonging from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Interpersonal Needs Questionnaire has a minimum possible score of 15, and maximum possible score of 105, wherein higher scores reflect higher perceived burdensomeness and thwarted belonging.
Change in relationship satisfaction from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Couples Satisfaction Index has a minimum possible score of 0, and maximum possible score of 161, wherein higher scores reflect higher relationship satisfaction.

OTHER OUTCOMES:
Expectations of Treatment | baseline
  The Credibility/Expectancy Questionnaire consists of 6 items rated on a 1-9 or a 0%-100% scale, wherein higher scores reflect higher treatment credibility and expectancy.
Satisfaction with Care | 13 weeks after baseline (post-treatment)
  The Client Satisfaction Questionnaire has a minimum possible score of 8, and a maximum possible score of 32, wherein higher scores reflect greater satisfaction with the intervention.
Change in relationship conflict from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Revised Conflict Tactics Scale consists of 20 items rated on a 0-7 scale, wherein higher scores reflect more conflict.
Change in severity of depression from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Patient Health Questionnaire-9 has a minimum possible score of 0 and a maximum possible score of 27, wherein higher scores reflect higher severity of depression.
Changes in Posttraumatic Stress Disorder severity from baseline | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  The Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) has a minimum possible score of 0 and a maximum possible score of 80, wherein higher scores reflect more severe posttraumatic stress disorder symptomatology.
Outpatient Engagement | Delivered at baseline, 7 weeks after baseline (mid-treatment), 13 weeks after baseline (post-treatment), and 25 weeks after baseline
  Outpatient engagement will be measured with the Cornell Services Index, which is an instrument that elicits information about the quantity and timing of inpatient and outpatient care (both mental health and non-mental health) as well as self-help groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra E Khalifian, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No